CLINICAL TRIAL: NCT03761537
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, Multi-centre, Phase 3 Trial Investigating the Efficacy, Safety, and Tolerability of Tralokinumab Administered in Combination With Topical Corticosteroids to Adult Subjects With Severe Atopic Dermatitis
Brief Title: Tralokinumab in Combination With Topical Corticosteroids in Subjects With Severe Atopic Dermatitis - ECZTRA 7
Acronym: ECZTRA 7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0162-1346
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tralokinumab + TCS (Experimental): 4 subcutaneous (SC) injections of tralokinumab 150 mg as a loading dose on Day 0, followed by 2 SC injections of tralokinumab 150 mg every 2 weeks (Q2W) regimen for 26 weeks. The last administration of the Investigational Medicinal Product (IMP) occurred at Week 24. From Day 0 to Week 24, a Topical corticosteroid (TCS) cream was dispensed to the participants at each IMP dosing visit (e.g., Q2W). Participants were instructed to treat active lesions as needed and to discontinue the TCS treatment when control was achieved.
  Interventions: Drug: Tralokinumab
- Placebo + TCS (Placebo Comparator): 4 subcutaneous (SC) injections of placebo as a loading dose on Day 0, followed by 2 SC injections of placebo every 2 weeks (Q2W) regimen for 26 weeks. The last administration of the Investigational Medicinal Product (IMP) occurred at Week 24. From Day 0 to Week 24, a Topical corticosteroid (TCS) cream was dispensed to the participants at each IMP dosing visit (e.g., Q2W). Participants were instructed to treat active lesions as needed and to discontinue the TCS treatment when control was achieved.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tralokinumab — Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous (SC) administration.
  Arms: Tralokinumab + TCS
Other: Placebo — Placebo contains the same excipients in the same concentration only lacking tralokinumab.
  Arms: Placebo + TCS

SUMMARY:
Primary objective:

To demonstrate that tralokinumab in combination with topical corticosteroids (TCS) is superior to placebo in combination with TCS in treating severe AD in subjects who are not adequately controlled with or have contraindications to oral cyclosporine A (CSA).

Secondary objectives:

To evaluate the efficacy of tralokinumab in combination with TCS on severity and extent of AD, itch, and health-related quality of life compared to placebo in combination with TCS.

To evaluate the safety of tralokinumab in combination with TCS when treating severe AD in subjects who are not adequately controlled with or have contraindications to oral CSA compared to placebo in combination with TCS.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 and above
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for AD
* History of AD for 1 year or more
* Subjects with a history within 1 year prior to screening of inadequate response to treatment with topical medications or subjects for whom topical treatments are otherwise medically inadvisable
* AD involvement of 10% (or more) body surface area at screening and baseline (visit 3) according to component A of SCORAD
* Documented history of either no previous CSA exposure and not currently a candidate for CSA treatment OR previous exposure to CSA in which case CSA treatment should not be continued or restarted
* Subjects must have applied a stable dose of emollient twice daily (or more, as needed) for at least 14 days before randomisation

Key Exclusion Criteria:

* Subjects for whom TCSs are medically inadvisable in the opinion of the investigator
* Use of tanning beds or phototherapy (NBUVB, UVB, UVA1, PUVA), within 6 weeks prior to randomisation
* Treatment with immunomodulatory medications or bleach baths within 4 weeks prior to randomisation
* Treatment with topical phosphodiesterase-4 (PDE-4) inhibitor within 2 weeks prior to randomisation
* Receipt of any marketed or investigational biologic agent (e.g. cell-depleting agents or dupilumab) within 6 months prior to randomisation or until cell counts return to normal, whichever is longer
* History of any active skin infection within 1 week prior to randomisation
* History of a clinically significant infection (systemic infection or serious skin infection requiring parenteral treatment) within 4 weeks prior to randomisation
* A helminth parasitic infection within 6 months prior to the date informed consent is obtained that has not been treated with, or has failed to respond to, standard of care therapy
* Tuberculosis requiring treatment within the 12 months prior to screening. Evaluation will be according to local guidelines as per local standard of care
* History of any known primary immunodeficiency disorder including a positive HIV test at screening, or the subject taking antiretroviral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (59):
- Belgium (9):
  - Leo Pharma Investigationel Site, Brussels
  - Leo Pharma Investigationel Site, Edegem
  - Leo Pharma Investigationel Site, Ghent
  - Leo Pharma Investigationel Site, Herstal
  - Leo Pharma Investigationel Site, Kortrijk
  - Leo Pharma Investigationel Site, Leuven
  - Leo Pharma Investigationel Site, Liège
  - Leo Pharma Investigationel Site, Loverval
  - Leo Pharma Investigationel Site, Maldegem
- Czechia (5):
  - Leo Pharma Investigationel Site, Karlovy Vary
  - Leo Pharma Investigationel Site, Kutná Hora
  - Leo Pharma Investigationel Site, Ostrava
  - Leo Pharma Investigationel Site, Pardubice
  - Leo Pharma Investigationel Site, Prague
- France (5):
  - Leo Pharma Investigationel Site, Grenoble
  - Leo Pharma Investigationel Site, Nice
  - Leo Pharma Investigationel Site, Paris
  - Leo Pharma Investigationel Site, Pierre-Bénite
  - Leo Pharma Investigationel Site, Valence
- Germany (15):
  - Leo Pharma Investigationel Site, Aachen
  - Leo Pharma Investigationel Site, Augsburg
  - Leo Pharma Investigationel Site, Bad Bentheim
  - Leo Pharma Investigationel Site, Berlin
  - Leo Pharma Investigationel Site, Dresden
  - Leo Pharma Investigationel Site, Dülmen
  - Leo Pharma Investigationel Site, Frankfurt
  - Leo Pharma Investigationel Site, Halle
  - Leo Pharma Investigationel Site, Hanover
  - Leo Pharma Investigationel Site, Jena
  - Leo Pharma Investigationel Site, Kiel
  - Leo Pharma Investigationel Site, Mainz
  - Leo Pharma Investigationel Site, München
  - Leo Pharma Investigationel Site, Osnabrück
  - Leo Pharma Investigationel Site, Selters
- Poland (11):
  - Leo Pharma Investigationel Site, Bialystok
  - Leo Pharma Investigationel Site, Bochnia
  - Leo Pharma Investigationel Site, Bydgoszcz
  - Leo Pharma Investigationel Site, Gdansk
  - Leo Pharma Investigationel Site, Krakow
  - Leo Pharma Investigationel Site, Lodz
  - Leo Pharma Investigationel Site, Lublin
  - Leo Pharma Investigationel Site, Poznan
  - Leo Pharma Investigationel Site, Rzeszów
  - Leo Pharma Investigationel Site, Warsaw
  - Leo Pharma Investigationel Site, Wroclaw
- Spain (8):
  - Leo Pharma Investigationel Site, Granada, Andalusia
  - Leo Pharma Investigationel Site, Alicante
  - Leo Pharma Investigationel Site, Barcelona
  - Leo Pharma Investigationel Site, Bilbao
  - Leo Pharma Investigationel Site, Córdoba
  - Leo Pharma Investigationel Site, Madrid
  - Leo Pharma Investigationel Site, Pamplona
  - Leo Pharma Investigationel Site, Seville
- United Kingdom (6):
  - Leo Pharma Investigationel Site, Bradford
  - Leo Pharma Investigationel Site, Cottingham
  - Leo Pharma Investigationel Site, Kirkcaldy
  - Leo Pharma Investigationel Site, London
  - Leo Pharma Investigationel Site, Southampton
  - Leo Pharma Investigationel Site, Wakefield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the participant gave informed consent, they went through a 2- to 6-week screening period. Eligibility was assessed at the (first) screening visit and on Day 0 (hereinafter "baseline") prior to randomisation.
Groups:
- Tralokinumab + TCS: Participants in the treatment period (Week 0 to Week 26) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants received a loading dose of 600 mg tralokinumab at baseline followed by a dose of 300 mg tralokinumab Q2W from Week 2. The last dose of IMP was administered at Week 24.
- Placebo + TCS: Participants in the treatment period (Week 0 to Week 26) treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants were administered placebo at baseline followed by administration of placebo every second week from Week 2. The last dose of IMP was administered at Week 24.
Period: Overall Study
Arm/Group | Tralokinumab + TCS | Placebo + TCS
Started | 140 | 137
Completed | 125 | 120
Not Completed | 15 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tralokinumab + TCS | Placebo + TCS | Total
Number analyzed (Participants) | 140 | 137 | 277
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 33.0 [25.5 to 47.0] | 34.0 [26.0 to 45.0] | 34.0 [26.0 to 45.0]
Age, Customized [Count of Participants; unit: Participants]
  18-64 | 134 | 131 | 265
  65-84 | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 54 | 112
  Male | 82 | 83 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 134 | 133 | 267
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 137 | 135 | 272
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 25 | 27 | 52
  Czechia | 14 | 12 | 26
  Poland | 34 | 43 | 77
  United Kingdom | 5 | 9 | 14
  France | 12 | 7 | 19
  Germany | 22 | 18 | 40
  Spain | 28 | 21 | 49
Age at onset of atopic dermatitis [Median (Inter-Quartile Range); unit: Years] — Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  Years
    number analyzed (Participants) | 140 | 136 | 276
    (all) | 2.5 [1.0 to 12.5] | 3.0 [1.0 to 17.0] | 3.0 [1.0 to 15.0]
Duration of atopic dermatitis [Median (Inter-Quartile Range); unit: Years] — Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  Years
    number analyzed (Participants) | 140 | 136 | 276
    (all) | 26.0 [18.0 to 35.0] | 25.0 [17.0 to 34.0] | 26.0 [18.0 to 34.5]
Body surface area with atopic dermatitis [Median (Inter-Quartile Range); unit: Percentage affected] | 52.0 [36.5 to 70.0] | 52.0 [35.0 to 70.0] | 52.0 [35.0 to 70.0]
Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — IGA is used to evaluate the severity of atopic dermatitis. It is a 5-point score ranging from 0 (clear) to 4 (severe). Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  Participants
    Moderate Disease: number analyzed (Participants) | 138 | 137 | 275
    Moderate Disease | 68 | 70 | 138
    Severe Disease: number analyzed (Participants) | 138 | 137 | 275
    Severe Disease | 70 | 67 | 137
Eczema Area and Severity Index (EASI) [Median (Inter-Quartile Range); unit: Units on a scale] — EASI is used to evaluate the extent and severity of atopic dermatitis. It is a composite score ranging from 0 to 72 with a higher score indicating a more extensive and/or severe condition. Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  Units on a scale
    number analyzed (Participants) | 138 | 137 | 275
    (all) | 28.60 [22.40 to 38.00] | 29.10 [22.80 to 40.15] | 28.80 [22.40 to 39.60]
Scoring Atopic Dermatitis (SCORAD) [Median (Inter-Quartile Range); unit: Units on a scale] — SCORAD is used to evaluate the extent and severity of atopic dermatitis as well as subjective symptoms. The score ranges from 0 to 103 with a higher score indicating a more extensive and/or severe condition. Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  Units on a scale
    number analyzed (Participants) | 138 | 137 | 275
    (all) | 69.20 [61.50 to 76.50] | 68.90 [61.20 to 81.00] | 69.10 [61.40 to 78.90]
Dermatology Life Quality Index (DLQI) [Median (Inter-Quartile Range); unit: Units on a scale] — DLQI is used by the participant to evaluate the impact of their condition on 10 different aspects of health-related quality of life (HRQoL) over the last week. Each item is scored on a 4-point Likert scale ranging from 0 (not at all/not relevant) to 3 (very much). The total score which is the sum of the 10 items ranges from 0 to 30, with a higher score indicating a poorer HRQoL. Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  Units on a scale
    number analyzed (Participants) | 137 | 134 | 271
    (all) | 16.00 [11.00 to 21.00] | 16.00 [11.00 to 21.00] | 16.00 [11.00 to 21.00]
Worst Daily Pruritus numeric rating scale (NRS) (weekly average) [Median (Inter-Quartile Range); unit: Units on a scale] — Worst Daily Pruritus NRS is used by the participant to evaluate their worst itch severity over the past 24 hours. The score ranges from 0 ('no itch') to 10 ('worst itch imaginable'). Population: The number of participants analysed is different from the number of participants randomised due to missing data.
  Units on a scale
    number analyzed (Participants) | 137 | 136 | 273
    (all) | 7.43 [6.43 to 8.29] | 7.50 [6.59 to 8.37] | 7.43 [6.57 to 8.29]

OUTCOME MEASURES:

1. Primary Outcome: At Least 75% Reduction in Eczema Area and Severity Index (EASI75) From Week 0 to Week 16
Description: EASI (Eczema Area and Severity Index) is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Time Frame: Week 0 to Week 16
Population: Full analysis set (FAS). Of the 277 participants randomised to initial treatment, 275 were treated. Therefore, the FAS consisted of 275 participants (138 participants in the tralokinumab+TCS group + 137 participants in the placebo+TCS group).
Measure: Number; unit: Percentage of responders
Groups:
- Tralokinumab+TCS: Participants in the initial treatment period (Week 0 to Week 16) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants received a loading dose of 600 mg tralokinumab at Week 0 followed by a dose of 300 mg tralokinumab Q2W from Week 2 to Week 16.
- Placebo+TCS: Participants in the initial treatment period (Week 0 to Week 16) treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants were administered placebo at Week 0 followed by administration of placebo every second week from Week 2 to Week 16.
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 138 | 137
Percentage of responders | 64.2 | 50.5
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Subjects who received rescue treatment or permanently discontinued IMP, without prior subject-onset of the COVID-19 pandemic (SOC19), were considered non-responders after the relevant event occurred. Any data from subjects who had SOC19 as their first prior intercurrent event (ICE) were multiple imputed (MI) assuming missing at random (MAR) following start of SOC19. Data missing prior to any ICE were handled as non-response, except data missing due to the pandemic, which was MI assuming MAR; Test type: Superiority — The null hypothesis of no difference between Tralokinumab+TCS and placebo+TCS was tested at a 5% significance level against the 2-sided alternative that there was a difference; p = 0.018, Mantel Haenszel — This endpoint was the first endpoint in the sequential testing hierarchy; Mantel-Haenszel (MH) test stratified by prior CSA use and baseline disease severity. MH risk differences and standard errors combined by Rubin's rule; Risk Difference (RD) = 14.1, 95% CI 2-sided [2.5 to 25.7]

2. Secondary Outcome: Reduction of Worst Daily Pruritus Numeric Rating Scale (NRS) (Weekly Average) of at Least 4 From Week 0 to Week 16
Description: Subjects will assess their worst itch severity over the past 24 hours using an 11-point NRS ('Worst Daily Pruritus NRS') with 0 indicating 'no itch' and 10 indicating 'worst itch imaginable'.
Time Frame: Week 0 to Week 16
Population: Participants in the full analysis set with a Worst Daily Pruritus NRS (weekly average) of at least 4 at baseline (Week 0).
Measure: Number; unit: Percentage of responders
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 134 | 135
Percentage of responders | 45.5 | 35.6
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.106, Mantel Haenszel — This endpoint was the second endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 9.7, 95% CI 2-sided [-2.0 to 21.4]

3. Secondary Outcome: Change in Scoring Atopic Dermatitis (SCORAD) From Week 0 to Week 16
Description: SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Time Frame: Week 0 to Week 16
Population: Full analysis set (FAS).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 138 | 137
Units on a scale | -42.7 (1.6) | -34.1 (1.6)
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; Data collected after permanent discontinuation of IMP, after initiation of rescue treatment, or after subject-onset of the COVID-19 pandemic will not be included in the analysis; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Repeated measurements model — This was the third endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; Treatment effect at each visit adjusted for baseline SCORAD interacting with each visit, prior CSA, and baseline disease severity (IGA 3 or 4); Difference = -8.6, 95% CI 2-sided [-13.0 to -4.2]

4. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Score From Week 0 to Week 16
Description: DLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on different aspects of their health-related quality of life (HRQoL) over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4-point Likert scale (0 = not at all ∕not relevant; 1 = a little; 2 = a lot; 3 = very much). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor HRQoL.
Time Frame: Week 0 to Week 16
Population: Full Set Analysis (FAS).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 137 | 134
Units on a scale | -11.2 (0.4) | -9.6 (0.4)
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.009, Repeated measurements model — This was the fourth endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; Treatment effect at each visit adjusted for baseline DLQI interacting with each visit, prior CSA, and baseline disease severity (IGA 3 or 4); Difference = -1.5, 95% CI 2-sided [-2.6 to -0.4]

5. Secondary Outcome: Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16
Description: IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Week 16
Population: Full analysis set (FAS).
Measure: Number; unit: Percentage of responders
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 138 | 137
Percentage of responders | 40.9 | 26.0
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.005, Mantel Haenszel — This endpoint was the fifth endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 15.6, 95% CI 2-sided [4.8 to 26.3]

6. Secondary Outcome: At Least 75% Reduction in Eczema Area and Severity Index (EASI75) From Week 0 to Week 26
Description: as for outcome 1
Time Frame: Week 0 to Week 26
Population: Full analysis set (FAS).
Measure: Number; unit: Percentage of responders
Groups:
- Tralokinumab: Participants in the treatment period (Week 0 to Week 26) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants received a loading dose of 600 mg tralokinumab at baseline followed by a dose of 300 mg tralokinumab Q2W from Week 2. The last dose of IMP was administered at Week 24.
- Placebo: Participants in the treatment period (Week 0 to Week 26) treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants were administered placebo at baseline followed by administration of placebo every second week from Week 2. The last dose of IMP was administered at Week 24.
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 138 | 137
Percentage of responders | 68.8 | 55.3
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.014, Mantel Haenszel — This endpoint was the sixth endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 14.1, 95% CI 2-sided [2.9 to 25.3]

7. Secondary Outcome: Reduction of Worst Daily Pruritus Numeric Rating Scale (NRS) (Weekly Average) of at Least 4 From Week 0 to Week 26
Description: Subjects will assess their worst itch severity over the past 24 hours using an 11-point numeric rating scale ('Worst Daily Pruritus NRS') with 0 indicating 'no itch' and 10 indicating 'worst itch imaginable'.
Time Frame: Week 0 to Week 26
Population: as for outcome 2
Measure: Number; unit: Percentage of responders
Groups:
- Tralokinumab+TCS: Participants in the treatment period (Week 0 to Week 26) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants received a loading dose of 600 mg tralokinumab at baseline followed by a dose of 300 mg tralokinumab Q2W from Week 2. The last dose of IMP was administered at Week 24.
- Placebo+TCS: Participants in the treatment period (Week 0 to Week 26) treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants were administered placebo at baseline followed by administration of placebo every second week from Week 2. The last dose of IMP was administered at Week 24.
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 134 | 135
Percentage of responders | 47.2 | 39.7
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.228, Mantel Haenszel — This endpoint was the seventh endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; HaenszMantelel (MH) test stratified by prior CSA use and baseline disease severity. MH risk differences and standard errors combined by Rubin's rule; Risk Difference (RD) = 7.3, 95% CI 2-sided [-4.6 to 19.2]

8. Secondary Outcome: Change in Scoring Atopic Dermatitis (SCORAD) From Week 0 to Week 26
Description: as for outcome 3
Time Frame: Week 0 to Week 26
Population: Full analysis set (FAS).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 138 | 137
Units on a scale | -46.3 (1.5) | -37.3 (1.6)
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Repeated measurements model — This endpoint was the eighth endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; Unstructured covariance matrix. Adjusted for baseline SCORAD in interaction with each visit, prior CSA use, and baseline disease severity (IGA 3 or 4); Difference = -8.9, 95% CI 2-sided [-13.2 to -4.6]

9. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Score From Week 0 to Week 26
Description: as for outcome 4
Time Frame: Week 0 to Week 26
Population: Full Set Analysis (FAS).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 137 | 134
Units on a scale | -11.5 (0.4) | -9.9 (0.4)
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.005, Repeated measurements model — This endpoint was the ninth endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; Unstructured covariance matrix. Adjusted for baseline DLQI in interaction with each visit, prior CSA use, and baseline disease severity (IGA 3 or 4); Difference = -1.6, 95% CI 2-sided [-2.7 to -0.5]

10. Secondary Outcome: Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 26
Description: as for outcome 5
Time Frame: Week 26
Population: Full analysis set (FAS).
Measure: Number; unit: Percentage of responders
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 138 | 137
Percentage of responders | 47.0 | 33.4
Statistical Analysis 1: Comparison: Tralokinumab+TCS vs Placebo+TCS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.014, Mantel Haenszel — This endpoint was the tenth endpoint in the sequential testing hierarchy. Acceptance of this endpoint depends on prior endpoints' acceptance; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 14.3, 95% CI 2-sided [2.9 to 25.6]

11. Secondary Outcome: Frequency of Anti-drug Antibodies (ADA) From Week 0 to Week 40
Description: Presence of ADA from Week 0 to Week 40 was measured. Data were reported in the following categories: positive (presence of ADA at baseline and/or presence of ADA at at least 1 post-baseline assessment), perishing (presence of ADA at baseline and absence of ADA at all post-baseline assessments), negative (absence of ADA at all assessments), no post-baseline ADA assessment.
Time Frame: Week 0 to Week 40
Measure: Count of Participants; unit: Participants
Groups:
- Tralokinumab+TCS; Placebo+TCS: Participants in the entire trial period, including the treatment period (Week 0 to Week 26) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed, and the safety follow-up period (up to Week 40).
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 138 | 137
Participants
  Positive | 2 | 3
  Negative | 134 | 133
  Perishing | 1 | 1
  No post-baseline ADA assessment | 1 | 0

12. Secondary Outcome: Number of Adverse Events From Week 0 to Week 40
Description: All adverse events are presented below under Adverse Events
Time Frame: Week 0 to Week 40
Measure: Number; unit: number of adverse events
Arm/Group | Tralokinumab+TCS | Placebo+TCS
Number analyzed (Participants) | 138 | 137
number of adverse events | 389 | 435

ADVERSE EVENTS:
Time Frame: Treatment period (Week 0 to Week 26), safety follow-up period (Week 26 to Week 40).
Description: The analysis was conducted based on the safety analysis set which consisted of subjects exposed to at least 1 dose of investigational medicinal product (IMP e.g., tralokinumab or placebo).
  In the category Other adverse events (AEs), all AEs will be reported in the safety follow-up period, whereas a frequency threshold at 2% AEs will apply for the treatment period, except that all AEs will be reported if also part of the safety follow-up period.
Groups:
- Treatment Period: Tralokinumab+TCS: Participants in the treatment period (Week 0 to Week 26) treated with tralokinumab every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants received a loading dose of 600 mg tralokinumab at baseline followed by a dose of 300 mg tralokinumab Q2W from Week 2. The last dose of IMP was administered at Week 24.
  For the treatment period, only AEs with a frequency above 2% will be reported. The exception is that AEs reported in the safety follow-up period will also be reported for the treatment period. The total AEs will represent all AEs reported in the treatment period.
- Treatment Period: Placebo+TCS: Participants in the treatment period (Week 0 to Week 26) treated with placebo every second week (Q2W) and topical corticosteroid (TCS) as needed.
  Participants were administered placebo at baseline followed by administration of placebo every second week from Week 2. The last dose of IMP was administered at Week 24.
  For the treatment period, only AEs with a frequency above 2% will be reported. The exception is that AEs reported in the safety follow-up period will also be reported for the treatment period. The total AEs will represent all AEs reported in the treatment period.
- Safety Follow-up Period: Tralokinumab+TCS; Safety Follow-up Period: Placebo+TCS: Participants who spent any amount of time in the safety follow-up period, independently of the treatment(s) received before. No treatment was administered to the participants during the safety follow-up period. Eligible participants were invited to enter a long-term extension trial conducted under a separate protocol (LP0162-1337, ECZTEND).
  For the safety follow-up period, all AEs will be reported.
Arm/Group | Treatment Period: Tralokinumab+TCS | Treatment Period: Placebo+TCS | Safety Follow-up Period: Tralokinumab+TCS | Safety Follow-up Period: Placebo+TCS
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/137 | 0/75 | 0/83
Serious Adverse Events (participants affected / at risk) | 1/138 | 5/137 | 0/75 | 1/83
Other Adverse Events (participants affected / at risk) | 107/138 | 108/137 | 4/75 | 6/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: Tralokinumab+TCS (N=138) | Treatment Period: Placebo+TCS (N=137) | Safety Follow-up Period: Tralokinumab+TCS (N=75) | Safety Follow-up Period: Placebo+TCS (N=83)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: Tralokinumab+TCS (N=138) | Treatment Period: Placebo+TCS (N=137) | Safety Follow-up Period: Tralokinumab+TCS (N=75) | Safety Follow-up Period: Placebo+TCS (N=83)
Viral upper respiratory tract infection (Infections and infestations) | 37 (53) | 35 (46) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (12) | 10 (11) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 6 (6) | 2 (3) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 5 (8) | 6 (6) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 5 (6) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (4) | 5 (5) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Dermatitis infected (Infections and infestations) | 2 (2) | 5 (10) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 (11) | 16 (26) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (12) | 5 (6) | 0 (0) | 0 (0)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 21 (25) | 13 (18) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 4 (5) | 1 (3) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (9) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (7) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (8) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 6 (8) | 5 (5) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 7 (7) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT03761537/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03761537/SAP_001.pdf